CLINICAL TRIAL: NCT06113367
Title: Carcinomes urothéliaux Des Voies excrétrices supérieures traitées en Vie réelle Par immunothérapie (VESUVIO) : étude rétrospective Nationale
Brief Title: Immunotherapy in Upper Tract Urothelial Carcinoma
Acronym: VESUVIO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230738
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with advanced/metastatic UTUC treated with second-line anti-PD-(L)1 immunotherapy
  Interventions: Other: Evaluation of anti-PD-(L)1 immunotherapy efficacy

INTERVENTIONS:
Other: Evaluation of anti-PD-(L)1 immunotherapy efficacy — Non Applicable, research on data

SUMMARY:
Upper-tract urothelial carcinoma (UTUC) is a rare tumor. Standard treatment of localized disease is most often radical nephroureterectomy.

In advanced/metastatic disease, treatments follow the standards for urothelial carcinoma including platinum-based chemotherapy and anti-PD(L)1 (Programmed death (ligand) 1) immunotherapy, with no regard as to the primary disease site (bladder or upper tract). Given the rarity of UTUC, efficacy data in the UTUC subgroup of advanced urothelial carcinoma is scarce.

UTUC show distinct pahological and molecular features, including higher prevalence of microsatellite instability and of abnormalities in the FGFR (fibroblast growth factor receptors) gene family. These specific features may impact outcomes of immunotherapy in advanced/metastatic UTUC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and more
* Diagnosis of urothelial carcinoma (with or without variant histology)
* Advanced/metastatic disease not amenable to local treatment with curative intent
* Treatment with an anti-PD-(L)1 monoclonal antibody initiated between 2016 and 2022

Exclusion Criteria:

* Patient's opposition to this research
* Urothelial carcinoma of bladder or urethral primary site
* Non-urothelial tumor
* Maintenance immunotherapy initiated without disease progression

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced/metastatic UTUC treated with second-line anti-PD-(L)1 immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival on anti-PD-(L)1 immunotherapy | 2 years after immunotherapy initiation

SECONDARY OUTCOMES:
Best Objective Radiologic Response | Up to 7 years maximum
  Evaluated by RECIST v1.1 The Response Evaluation Criteria in Solid Tumors (RECIST) is a standard system to measure how cancer responds to different treatments.It permits to evaluate the response according to the evolution of the lesions.
Overall survival | 5 years after immunotherapy initiation
Progression free survival | 6 months after immunotherapy initiation
Progression free survival | 1 year after immunotherapy initiation
Progression free survival | 2 years after immunotherapy initiation
Progression free survival | 3 years after immunotherapy initiation
Duration of immunotherapy treatment | Up to 7 years after immunotherapy initiation
  Treatment tolerability
Reasons for treatment discontinuation | Up to 7 years after immunotherapy initiation
Translational study of predictive biomarkers of efficacy | Up to 7 years after immunotherapy initiation

IPD SHARING:
Plan to Share IPD: Undecided